CLINICAL TRIAL: NCT06549452
Title: MhOVE-PPH Study: Mobile Health Intervention to Improve Exercise in Pediatric PH
Brief Title: Mobile Health Intervention to Improve Exercise in Pediatric PH
Acronym: MhOVE-PPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of California, San Francisco (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Eric Austin, Director, Vanderbilt Pediatric Pulmonary Hypertension Program (Allergy/Immunology/Pulmonary Medicine) and Associate Professor of Pediatrics (Allergy/Immunology/Pulmonary Medicine), Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 240771; 1R34HL173389 (NIH)
Record Dates: First submitted 2024-06-24; First posted 2024-08-12 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized, un-blinded, parallel group, Phase II study of 50 subjects with PAH. Eligible subjects will be randomly assigned to receive the mHealth intervention or usual care for twelve weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mHealth Intervention (Active Comparator): Patients will be randomized to the mHealth texting platform, which are messages designed to facilitate self-awareness, reinforce step targets, and link physical activity with a reward or memorable cue.
  Interventions: Device: mHealth Intervention
- Usual Care (Other): Routine medical care
  Interventions: Device: Usual Care

INTERVENTIONS:
Device: mHealth Intervention — Our HIPPA-compliant texting platform is linked to the Fitabase Interface. Real time activity data are transmitted from the participant's smartphone to Fitabase via cellular network. Participants will receive 3-5 texts/day in sync with their preferred schedule defined at enrollment and taking into account school schedules as relevant. These texts use personal, disease-specific, and provider information to deliver two types of messages customized to the current step count and sent in equal proportion. Messages are designed to facilitate self-awareness, reinforce step targets, and link physical activity with a reward or memorable cue.
  Arms: mHealth Intervention
Device: Usual Care — Routine medical care
  Arms: Usual Care

SUMMARY:
Children and adults with pulmonary arterial hypertension (PAH) have severely reduced daily activity compared to healthy populations. In adults, investigators recently demonstrated that lower baseline daily step counts associated with increased risk of hospitalization and worsening WHO functional class; similarly, reduced step counts associate with hospitalization in children with PAH. This application builds on our recently completed NIH-funded pilot mobile health (mHealth) trial in adult patients with PAH which demonstrated the ability to remotely increase step counts. The investigators now aim to: (1) adapt our mHealth intervention to the developmental needs and interests of adolescents; and, (2) determine if our intervention increases step counts in adolescents, providing the foundation for a larger trial to assess the impact on quality of life and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between ages 13-19 years.
* Diagnosed with idiopathic, heritable, or associated (connective tissue disease, drugs, or toxins) pulmonary arterial hypertension (PAH), or PAH due to simple congenital heart disease (i.e. atrial septal defect).
* WHO functional class I-III
* Stable PAH-specific medication regimen for three months prior to enrollment. Subjects with only a single diuretic adjustment in the prior three months will be included. Adjustments in IV prostacyclin for side effect management are allowed.
* Forced vital capacity >65% predicted with no or minimal interstitial lung disease based on reviews of imaging studies by PI and medical monitor.

Exclusion Criteria:

* Prohibited from normal activity due to wheelchair bound status, bed bound status, reliance on a cane/walker, activity-limiting angina, activity-limiting osteoarthritis, or other condition that limits activity.
* Pregnancy
* Diagnosis of PAH etiology other than idiopathic, heritable, or associated.
* Functional class IV heart failure
* Requirement of > 2 diuretic adjustment in the prior three months.
* Preferred form of activity is not measured by an activity tracker (swimming, yoga, ice skating, stair master, or activities on wheels such as bicycling or rollerblading).
* Involved in any other investigational intervention.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in average daily step count from baseline to 12 weeks | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on average daily step count from baseline to 12 weeks.
  Accelerometry is a direct measure of physical activity in patients' day-to-day lives. Step counts will be measured using the Fitbit device monitor, a lightweight device that has a three-axis acceleration sensor, altimeter, vibration motor, and optical heart rate monitor.

SECONDARY OUTCOMES:
Change in Quality of Life as measured by the Short Form 36-Item Health Survey (SF-36) | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on quality of life between baseline and Week 12.
  The SF36 is one of the most widely used generic measures of subjective health status. The SF36 includes one multi-item scale that assesses eight health concepts.
  Scoring the SF 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per a scoring key. All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the low
Change in Quality of Life as measured by the emPHasis-10 | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on quality of life between baseline and Week 12.
  The emPHasis-10 is a pulmonary hypertension-specific questionnaire to assess health related quality of life. It covers breathlessness, fatigue and lack of energy, social restrictions, and concerns regarding effects on patient's significant others, such as family and friends. Each item is scored on a semantic differential six-point scale (0-5), with contrasting adjectives at each end. A total emPHasis-10 score is derived using simple aggregation of the 10 items. emPHasis-10 scores range from 0 to 50, higher scores indicate worse quality of life.
Change in Quality of Life as measured by the Pediatric Quality of Life Inventory (PedsQL) | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on quality of life between baseline and Week 12.
  The Pediatric Quality of Life Inventory (PedsQL) Measurement Model is a modular approach to measuring health-related quality of life (HRQOL) in healthy children and adolescents and those with acute and chronic health conditions. The PedsQL integrates seamlessly both generic core scales and disease-specific modules into one measurement system, which generally takes about 4 minutes to complete. Each item is scored on a 5-point Likert scale from 0 (Never) to 4 (Almost always), then reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Higher scores indicate better health-related quality of life.
Change in Quality of Life as measured by the Pediatric Inventory for Parents (PIP) | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on quality of life between baseline and Week 12.
  The PIP is a questionnaire comprising 42 items, grouped into four domains or subscales: medical care, communication, emotional functioning, and role function. Its purpose is to measure the levels of stress suffered by parents caring for a child with a chronic disease. Responses are provided using a five-point Likert scale, ranging from 1 ("never/not at all") to 5 ("very often/extremely"). Higher scores indicate higher levels of stress.
Difference in total daily activity from baseline to 12 weeks | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on total daily activity time from baseline to 12 weeks. Activity time is defined as time spent above 3 metabolic equivalents.
  Accelerometry is a direct measure of physical activity in patients' day-to-day lives. Activity time will be measured using the Fitbit device monitor, a lightweight device that has a three-axis acceleration sensor, altimeter, vibration motor, and optical heart rate monitor.
Difference in unadjusted raw daily steps from baseline to 12 weeks | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on unadjusted change in raw daily steps from baseline to 12 weeks.
  Accelerometry is a direct measure of physical activity in patients' day-to-day lives. Step counts and will be measured using the Fitbit device monitor, a lightweight device that has a three-axis acceleration sensor, altimeter, vibration motor, and optical heart rate monitor.
Difference in total daily aerobic time from baseline to 12 weeks | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on total daily aerobic time from baseline to 12 weeks. Aerobic time is defined as the total time spent walking continuously for > 10 minutes without breaking for > 1 minute.
  Accelerometry is a direct measure of physical activity in patients' day-to-day lives. Aerobic time will be measured using the Fitbit device monitor, a lightweight device that has a three-axis acceleration sensor, altimeter, vibration motor, and optical heart rate monitor.
Difference in frequency of goal attainment from baseline to 12 weeks | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on frequency (% days) of goal attainment from baseline to 12 weeks.
  Accelerometry is a direct measure of physical activity in patients' day-to-day lives. Frequency (% days) of goal attainment will be measured using the Fitbit device monitor, a lightweight device that has a three-axis acceleration sensor, altimeter, vibration motor, and optical heart rate monitor.
Difference in mean daily steps during week 12 and week 18 | Week 12 & Week 18
  To assess the effect of a mHealth intervention or no intervention on mean daily steps during week 12 and week 18.
  Accelerometry is a direct measure of physical activity in patients' day-to-day lives. Step counts will be measured using the Fitbit device monitor, a lightweight device that has a three-axis acceleration sensor, altimeter, vibration motor, and optical heart rate monitor.
Difference in B-type natriuretic peptide levels from baseline to 12 weeks | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on B-type natriuretic peptide levels (pg/mL) between baseline and 12 weeks.
Difference in 6-Minute walk test distance from baseline to 12 weeks | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on the 6-minute walk test distance (meters) between baseline and 12 weeks.
Difference in Echocardiographic pericardial effusion from baseline to 12 weeks | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on Echocardiographic pericardial effusion from baseline to 12 weeks.
Difference in Echocardiographic maximal tricuspid regurgitant velocity from baseline to 12 weeks | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on Echocardiographic maximal tricuspid regurgitant velocity from baseline to 12 weeks.
Difference in Echocardiographic measurement of RV fractional area change (FAC) from baseline to 12 weeks | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on Echocardiographic measurement of RV fractional area change (FAC) from baseline to 12 weeks.
Time to clinical worsening | Baseline to 12 weeks
  To assess the effect of a mHealth intervention or no intervention on a composite outcome of PAH-related hospitalization, medication regimen escalation, decrease in vital status, and all-cause mortality at 12 weeks after randomization. Clinical worsening events are defined as death (all causes), hospitalizations due to worsening pulmonary arterial hypertension (PAH), escalation in WHO functional class, and initiation of an inhaled or infused prostacyclin (PGI2) for the treatment of worsening PAH.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Austin, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No